CLINICAL TRIAL: NCT04635059
Title: Pacritinib for Biochemical Relapse After Definitive Treatment for Prostate Cancer
Acronym: BLAST
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: futility and drug supplier in favor of new metastatic protocol.
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Deepak Kilari, Associate Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00040162
Record Dates: First submitted 2020-11-04; First posted 2020-11-18 (Actual); Results first posted 2024-12-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pacritinib (Experimental): Pacritinib is an oral drug.
  Interventions: Drug: Pacritinib

INTERVENTIONS:
Drug: Pacritinib — Pacritinib is an oral drug which will be taken daily on a 28-day cycle at a dose of 200 mg twice a day (BID).
  Other Names: SB1518

SUMMARY:
This is a single-arm, open-label study using pacritinib for patients with histologically confirmed prostate adenocarcinoma, status post definitive treatment and biochemical recurrence.

DETAILED DESCRIPTION:
This phase 2, single-arm, open-label study using pacritinib will treat patients with histologically confirmed prostate adenocarcinoma, status post definitive treatment and biochemical recurrence.

The primary objective of this study is to determine the effect of pacritinib on the time to prostate-specific antigen (PSA) progression in patients with biochemical relapse of prostate cancer (defined as the length of time that a given subject will be alive and free from PSA progression per Prostate Cancer Working Group 3 (PCWG3) guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 years.
2. Histologically or cytologically confirmed prostate adenocarcinoma.
3. Prior radical prostatectomy or definitive radiation.
4. Biochemically recurrent prostate cancer with PSA doubling time ≤ 9 months at the time of study entry (calculated per Memorial Sloan Kettering Cancer Center (MSKCC) prostate nomogram: https://www.mskcc.org/nomograms/prostate/psa_doubling_time). Calculation of PSA doubling time should include the use of all available PSA values obtained within the past 12 months prior to randomization, with a minimum of three values separated by at least two weeks apart. The PSA values used to calculate the PSA doubling time must all be ≥ 0.1 ng/mL and should be measured in the same laboratory whenever feasible.
5. Prior adjuvant or salvage radiation or not a candidate for radiation based upon clinical assessment of disease characteristics and patient comorbidities. (N/A for patients who underwent definitive radiation therapy).
6. Screening PSA > 0.5 ng/mL.
7. No definitive evidence of metastases on screening computerized tomography scan (CT) or magnetic resonance imaging (MRI) of abdomen/pelvis and radionuclide whole-body bone scan per the judgment of the investigator. Abdominal and/or pelvic lymph nodes measuring 1.5 cm or less in short axis diameter are allowed. Lesions identified on other imaging modalities (e.g. prostate specific membrane antigen (PSMA) or choline positron emission tomography (PET)) that are not visualized on CT and/or MRI or radionuclide bone scan are allowed. Equivocal lesions on bone scan should be followed up with additional imaging as clinically indicated.
8. Screening serum testosterone > 150 ng/dL.
9. Eastern Cooperative Oncology Group (ECOG) Performance Status grade 0 or 1 or Karnofsky Performance Status ≥ 70.
10. No prior Janus Kinase 2 (JAK2) inhibitor treatment.
11. Male patients, even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following:

    • Practice effective barrier contraception during the entire study period and through 60 calendar days after the last dose of study agent
12. Ability to understand a written informed consent document, and the willingness to sign it.
13. Left ventricular cardiac ejection fraction of ≥50% by echocardiogram or multigated acquisition (MUGA) scan.
14. Willing to provide blood and tissue for research analysis. (encouraged but not necessary for inclusion in trial).
15. Adequate organ function as defined by the following laboratory values at screening:

    * Serum aspartate transaminase (AST), serum glutamic oxaloacetic transaminase (SGOT) and serum alanine transaminase (ALT), serum glutamic pyruvic transaminase (SGPT) < 2.5 x upper limit of normal (ULN).
    * Total serum bilirubin ≤1.5 x ULN. In subjects with Gilbert's syndrome, if total bilirubin is >1.5 × ULN, measure direct and indirect bilirubin and if direct bilirubin is ≤1.5 × ULN, the subject may be eligible).
    * Serum potassium ≥ 3.5 mmol/L. Supplementation and re-screening is allowed.
    * Estimated glomerular filtration rate (GFR) > 45 ml/min using Cockroft-Gault equation.
    * Platelets ≥ 100,000/mL independent of transfusion and/or growth factors within three months prior to randomization.
    * Hemoglobin ≥ 9.0 g/dL independent of transfusion and/or growth factors within three months prior to randomization.
    * Absolute neutrophil count ≥500/µL.
    * Serum albumin ≥ 3.0 g/dL.
    * Adequate coagulation defined by prothrombin time (PT) / international normalized ratio (INR) and partial thromboplastin time (PTT) ≤ 1x.5 ULN.

Exclusion Criteria:

1. Previously treated with pacritinib.
2. Prior systemic treatment with androgen deprivation therapy and/or first-generation anti-androgen (e.g. bicalutamide, nilutamide, flutamide) for biochemically recurrent prostate cancer. Prior androgen deprivation therapy (ADT) and/or first-generation anti-androgen in the (neo)adjuvant, definitive and/or salvage setting in conjunction with radiation or surgery is allowed provided last effective dose of ADT and/or first-generation anti-androgen is > 9 months prior to the date of randomization and the total duration of prior therapy is ≤ 36 months.
3. Prior treatment with 17α-hydroxy / 17,20-lyase (CYP17) inhibitor (e.g., ketoconazole, abiraterone acetate, galeterone) or next-generation androgen receptor antagonist including apalutamide or enzalutamide.
4. Prior chemotherapy for prostate cancer except if administered in the neoadjuvant or adjuvant setting and last dose <= 6 months from randomization.
5. Use of 5-alpha reductase inhibitor within 42 days prior to randomization.
6. Use of investigational agents within 28 days prior to randomization.
7. Use of other prohibited medications within seven days prior to Cycle 1 Day 1 on study (see Appendix 3 and 4 for list of prohibited medications).
8. Systemic treatment with a strong Cytochrome P450 3A4 (CYP3A4) inhibitor or a strong cytochromes P450 (CYP450) inducer within 14 days prior to treatment Day 1.
9. Prior bilateral orchiectomy.
10. Uncontrolled hypertension.
11. Baseline severe hepatic impairment (Child-Pugh Class B & C).
12. An intercurrent illness that is not controlled, such as active infection, psychiatric illness/social situations that would limit compliance with study requirements.
13. Any chronic medical condition requiring a higher dose of corticosteroid than an equivalent of 10 mg prednisone/prednisolone per day.
14. Significant recent bleeding history, as defined as National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade≥2 within three months prior to treatment Day 1, unless precipitated by an inciting event (e.g., surgery, trauma, or injury)
15. Systemic treatment with medications that increase the risk of bleeding, including anticoagulants (warfarin, direct oral anticoagulant, etc.), antiplatelet agents (except for aspirin dosages of ≤ 100mg/day), vascular endothelial growth factor (anti-VEGF) agents, and daily use of COX-1 inhibiting nonsteroidal anti-inflammatory agents (NSAIDs) within 14 days prior to treatment Day 1.
16. Systemic treatment with medications that can prolong the time from the start of the Q wave to the end of the T wave (QT interval) within 14 days prior to treatment Day 1. Shorter washout periods may be permitted with the approval of the principal incestigator, provided that the washout period is at least five half-lives of the drug prior to treatment Day 1.
17. Any history of CTCAE grade ≥2 cardiac conditions within six months before treatment Day 1. Patients with asymptomatic grade 2 non-dysrhythmia cardiovascular conditions may be considered for inclusion, with the approval of the PI, if stable and unlikely to affect patient safety.
18. QT corrected by the Fridericia method (QTcF) prolongation >450 ms or other factors that increase the risk for QT interval prolongation (e.g., heart failure, hypokalemia [defined as serum potassium <3.0 mEq/L that is persistent and refractory to correction]), or history of long QT interval syndrome.
19. New York Heart Association Class II, III, or IV congestive heart failure (Appendix 7).
20. Any active gastrointestinal (GI) or metabolic condition that could interfere with absorption of oral medication.
21. Active or uncontrolled inflammatory or chronic functional bowel disorder such as Crohn's disease, inflammatory bowel disease, chronic diarrhea, or chronic constipation.
22. Other malignancy within three years prior to treatment Day 1, other than curatively treated basal cell or squamous cell skin or corneal cancer; curatively treated carcinoma in situ of the cervix; or in situ breast carcinoma after complete surgical resection.
23. Uncontrolled intercurrent illness, including, but not limited to, ongoing active infection, psychiatric illness, or social situation that, in the judgment of the treating physician, would limit compliance with study requirements.
24. Known seropositivity for human immunodeficiency virus.
25. Known active hepatitis A, B, or C virus infection.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Kilari, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pacritinib
Started | 6
Completed | 2
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Pacritinib
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients With Six-month PSA Progression-free Survival.
Description: PSA progression-free survival is defined as the length of time that a subject will be alive and free from PSA progression per PCWG3 guidelines.
Time Frame: Six months
Measure: Count of Participants; unit: Participants
Arm/Group | Pacritinib
Number analyzed (Participants) | 6
Participants | 0

2. Secondary Outcome: PSA Levels
Description: PSA level in blood is measured in units of nanograms per milliliter.
Time Frame: Cycle1Day1 (month 0), every month up to month 4.
Population: Two subjects were not tested in month 4.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pacritinib
Number analyzed (Participants) | 6
ng/mL
  PSA at C1D1 (month 0), ng/mL | 1.9 (.5)
  PSA at month 1, ng/mL | 3.2 (.8)
  PSA at month 2, ng/mL | 4.1 (1.3)
  PSA at month 3, ng/mL | 4.7 (.8)
  PSA at month 4, ng/mL: number analyzed (Participants) | 4
  PSA at month 4, ng/mL | 5.7 (.3)

3. Secondary Outcome: Testosterone Measurement
Description: Serum testosterone will be measured in nanograms per deciliter.
Time Frame: Baseline and three months
Population: Two subjects were not tested in month 3.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Pacritinib
Number analyzed (Participants) | 6
ng/dL
  Testosterone at screening, ng/dL | 390 (280)
  Testosterone at 3 months, ng/dL: number analyzed (Participants) | 4
  Testosterone at 3 months, ng/dL | 330 (181)

ADVERSE EVENTS:
Time Frame: 2 Years
Arm/Group | Pacritinib
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pacritinib (N=6)
Alanine aminotransferase increased (Investigations) | 1 (2)
Alkaline phosphatase increased (Investigations) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Belching (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Heavy eyelids (Eye disorders) | 1 (1)
Fatigue (General disorders) | 6 (6)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyperlipidemia (Metabolism and nutrition disorders) | 5 (5)
Hypertension (Vascular disorders) | 6 (6)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Salivary duct inflammation (Gastrointestinal disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 (2)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Testosterone deficiency (Endocrine disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 3 (3)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/59/NCT04635059/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-22): https://cdn.clinicaltrials.gov/large-docs/59/NCT04635059/ICF_001.pdf